CLINICAL TRIAL: NCT02143141
Title: Eliminating Long Acting Spinal Narcotic Use and Its Associated Side Effects for Those Who do Not Need it After Cesarean Delivery
Brief Title: Low Pain Prediction in Cesarean Section Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: feasibility of population needed to complete study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00017294
Record Dates: First submitted 2014-03-27; First posted 2014-05-20 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Scheduled Cesarean Sections; Postoperative Pain Management; Side Effects
Keywords: postoperative pain; narcotic side effects
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- duramorph (Active Comparator): duramorph 150 mcg administered spinally with placebo capsules administered by mouth every 6 hours x 4 doses during first 24 hours
  Interventions: Drug: duramorph
- no duramorph (Experimental): no duramorph is administered spinally for surgery; subjects receive acetaminophen 1 G orally x 4 doses during first 24 hours postoperatively
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: duramorph — duramorph 150 mcg given with spinal anesthetic, then receipt of placebo capsules postoperatively. evaluation postoperative day 1 for measurement of itching, nausea, vomiting, pain and itching.
  Other Names: duramorph versus placebo
  Arms: duramorph
Drug: placebo — placebo in an equal volume to that of duramorph 150 mcg given with spinal anesthetic, then receipt of oral acetaminophen 1000mg during first 24 hours postoperatively. evaluation postoperative day 1 for measurement of itching, nausea, vomiting, pain and itching.
  Arms: no duramorph

SUMMARY:
The investigators are attempting to see if eliminating the amount of long acting spinal narcotic during cesarean section delivery will demonstrate pain scores with movement when evaluated 24 hours postoperatively as those that receive the standard dosage of spinal narcotic when combined with oral acetaminophen or placebo. The investigators also are evaluating if there are decreased side effects related to decreased narcotic usage.

DETAILED DESCRIPTION:
Subjects are randomized on the morning of surgery to receive a standard dose of spinal narcotic or to receive no long acting spinal narcotic. The subjects may or may not also receive acetaminophen orally postoperatively. Pain scores are done on postoperative day one as well as evaluation of potential narcotic side effects such as nausea/vomiting, itching, and sedation.

ELIGIBILITY:
Inclusion Criteria:

* anticipated pain level estimated to be in the lowest 20th percentile (calculated <34.3 utilizing our standard preoperative questionnaire)
* age >/= 18
* not allergic to any study medications to be utilized in this study
* singleton pregnancy

Exclusion Criteria:

* allergies to morphine or acetaminophen
* diagnosis of a chronic pain disorder
* weight >300 lbs
* hepatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Booth, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment occurred between December 2011 and September 2013. The study was terminated due to extreme difficulty in recruiting patients willing to participate in the study.
Period: Overall Study
Arm/Group | Duramorph | no Duramorph
Started | 7 | 6
Completed | 6 | 6
Not Completed | 1 | 0
Not completed — pain scores at 24 hours not collected | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duramorph | no Duramorph | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Full Range); unit: years] | 32 [27 to 35] | 30 [21 to 36] | 31 [21 to 36]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female participants | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 13
gravida [Mean (Full Range); unit: number] — number of times a woman has been pregnant
  number | 3 [2 to 5] | 2 [1 to 4] | 2 [1 to 5]
para [Mean (Full Range); unit: number] — number of births a woman has had after 20 weeks of gestation
  number | 1 [1 to 2] | 1 [0 to 2] | 1 [0 to 2]
estimated gestational age of fetus [Mean (Full Range); unit: weeks] | 39 [39 to 40] | 39 [39 to 40] | 39 [39 to 40]
height [Mean (Full Range); unit: inches] | 64.8 [63 to 68] | 64.5 [62 to 69] | 64.6 [62 to 69]
weight [Mean (Full Range); unit: pounds] | 206 [160 to 267] | 166 [130 to 214] | 186 [130 to 267]

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain assessment is made using a Visual Analog Scale (VAS). VAS is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Scale ranges from 0 indicating no pain to 100 indicating the most severe pain.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duramorph | no Duramorph
Number analyzed (Participants) | 7 | 6
units on a scale | 56 (27) | 21 (11)

2. Secondary Outcome: Itching
Description: The itching assessment is made using a Visual Analog Scale (VAS). VAS is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Scale ranges from 0 indicating no itching to 100 indicating the most severe itching.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duramorph | no Duramorph
Number analyzed (Participants) | 7 | 6
units on a scale | 55.3 (21.7) | 1.3 (3.3)

3. Secondary Outcome: Nausea/Vomiting
Description: The nausea/vomiting assessment is made using a Visual Analog Scale (VAS). VAS is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. Scale ranges from 0 indicating no nausea/vomiting to 100 indicating the most severe nausea/vomiting.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duramorph | no Duramorph
Number analyzed (Participants) | 7 | 6
units on a scale | 37 (38.2) | 6.2 (15.1)

ADVERSE EVENTS:
Arm/Group | Duramorph | no Duramorph
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed. Extreme difficulty in recruiting participants to participate in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No